CLINICAL TRIAL: NCT03986424
Title: Multi-center Open Comparative Randomized Study of Efficacy and Safety of Akatinol Memantine 20 mg (Single-doses) vs. Akatinol Memantine 10 mg (Double-doses) in Patients With Moderate and Moderately Severe Vascular Dementia
Brief Title: Local Study of Akatinol Memantine in VaD in Russia
Acronym: MIND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Collaborators: LLC Merz Pharma, Russia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M900011005
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Vascular Dementia
MeSH Terms: conditions — Dementia, Vascular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Akatinol Memantine 20 mg (Experimental): Akatinol Memantine 20 mg once daily
  Interventions: Drug: Akatinol Memantine 20 mg
- Akatinol Memantine 10 mg (Active Comparator): Akatinol Memantine 10 mg twice daily
  Interventions: Drug: Akatinol Memantine 10 mg

INTERVENTIONS:
Drug: Akatinol Memantine 20 mg — Akatinol Memantine 20 mg to be taken orally, once daily, in the same time of the day
  Arms: Akatinol Memantine 20 mg
Drug: Akatinol Memantine 10 mg — Akatinol Memantine 10 mg to be taken orally, twice daily
  Arms: Akatinol Memantine 10 mg

SUMMARY:
The study evaluates the clinical efficacy and safety of Akatinol Memantine 20 mg (single-doses) vs. Akatinol Memantine 10 mg (double-doses) in patients suffering from moderate and moderately severe vascular dementia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient or his/her legal representative if the patient is declared incapable by a court decision.
* Understanding of study procedures and willingness to abide to all procedures during the course of the study by the patient or his/her legal representative.
* Male and female patients from 50 to 85 years of age (inclusive) suffering from moderate and moderately severe vascular dementia.
* Mini-Mental State Examination (MMSE) Test total scores of 10 to 20.
* Hachinski's Ischemic Score (HIS) of 7 or higher point.
* Availability in the anamnesis of instrumental confirmation of the diagnosis (data methods of neurovisualization - CT or MRT).
* For females: menopause or inability to conceive due to other reasons (hysterectomy, etc.).
* Availability of a relative or legal representative who lives with the patient, monitors him/her and cares for the patient.

Exclusion Criteria:

* Alzheimer's disease or secondary types of dementia.
* Epilepsy, seizures, schizophrenia, other psychoses, bipolar disorder, alcoholism, drug abuse (including the history thereof).
* Other clinically significant neurological or psychiatric disorders.
* Severe depression (Hamilton score, HAM-D > 18 points).
* Severe, unstable or decompensated physical disease (including clinically significant laboratory abnormalities) potentially affecting the trial findings.
* Contraindications to oral drug intake during the time period determined by the study protocol.
* Known hypersensitivity to the investigational product or any of its ingredients.
* Administration of nootropic, anti-dementia and typical antipsychotic drugs, tricyclic antidepressants, long-acting benzodiazepines, NMDA receptor antagonists (amantadine, ketamine, dextromethorphan) for 1 month before the enrollment and during the study.
* For females: pregnancy and breastfeeding.
* Evidence or suspicion that the patient might not comply with the study directive.
* Any reason or contraindication which in the investigator's opinion precludes participation in the study.
* Patient is direct relative of an employee of the study site or Merz Pharma LLC.
* Previous participation in this clinical study.
* Participation in another clinical trial within the last 12 weeks prior to screening or ongoing participation in a study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total ADAS-cog score points | 24 weeks
  ADAS-cog - Alzheimer's Disease Assessment scale, cognitive subscale

CONTACTS AND LOCATIONS:
Overall Officials: Merz Russia Medical Expert, Study Director — Merz Russia
Locations (4):
- Russia (4):
  - Federal State Budgetary Scientific Institution "Mental Health Research Center", Moscow
  - Federal State Autonomous Institution of Higher Learning "Peoples' Friendship University of Russia", Medical Institute, Moscow
  - Scientific Research Institute of Neurology, Merz Investigational Site #0070008, Moscow
  - Federal state budgetary military educational institution of higher education "Military Medical Academy named after S.M. Kirov" of the Ministry of defence of the Russian Federation, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No